CLINICAL TRIAL: NCT06316570
Title: Efficacy and Safety of Ticagrelor With Aspirin Dual Antiplatelet Therapy Combined With Intravenous Thrombolysis in Patients With Ischemic Stroke (TAPIS): a Multicenter, Randomized, Double-blind, Placebo-parallel Controlled Trial
Brief Title: Ticagrelor With Aspirin Dual Antiplatelet Therapy Combined With Intravenous Thrombolysis for Ischemic Stroke
Acronym: TAPIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, yilong Wang, Vice President of Beijing Tiantan Hospital, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HX-A-2023044; SF 2024-2-2045 (Other Grant/Funding Number: Capital health development research project)
Record Dates: First submitted 2024-03-12; First posted 2024-03-18 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Ischemic Stroke, Acute
Keywords: Ischemic Stroke; Antiplatelet Therapy; Intravenous Thrombolysis; Randomized Controlled Trial; Double Blind Study; Multicenter Study; Clinical Trial
MeSH Terms: conditions — Ischemic Stroke | interventions — Ticagrelor; Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual Antiplatelet Therapy (Experimental): This group will receive early dual antiplatelet therapy (Ticagrelor with Aspirin) combined with intravenous thrombolysis within 6 hours of the onset.
  Interventions: Drug: Early Dual Antiplatelet Therapy
- Placebo (Placebo Comparator): This group will receive placebo treatment (with same form and dosage) combined with intravenous thrombolysis within 6 hours of the onset.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Early Dual Antiplatelet Therapy — Day 1(within 6.0 hours of onset, before or after intravenous thrombolysis) : Ticagrelor (180mg) + Aspirin (100mg), one dose;
  Days 2-7: Ticagrelor (90mg/time, twice/day) + open-label Aspirin (100mg/time, once/day) ;
  Days 8-90: open-label Aspirin (100mg/time, once/day).
  Other Names: Ticagrelor and Aspirin
  Arms: Dual Antiplatelet Therapy
Drug: Placebo — Day 1(within 6.0 hours of onset, before or after intravenous thrombolysis) : Placebo of Ticagrelor (180mg) + Placebo of Aspirin (100mg), one dose;
  Days 2-7: Placebo of Ticagrelor (90mg/time, twice/day) + open-label Aspirin (100mg/time, once/day) ;
  Days 8-90: open-label Aspirin (100mg/time, once/day).
  Other Names: Placebo of Ticagrelor and Aspirin
  Arms: Placebo

SUMMARY:
Early antiplatelet therapy is promising for further improvement of functional prognosis on the basis of intravenous thrombolytic therapy. The primary purpose of this multicenter, randomized, double-blind, placebo-parallel controlled trial is to evaluate the efficacy and safety of the early dual antiplatelet therapy (within 6 hours of onset ) of ticagrelor with aspirin combined with intravenous thrombolysis in improving good functional outcome (mRS score 0-1) at 90 days inpatients with ischemic stroke.

DETAILED DESCRIPTION:
Theoretically, early administration of antiplatelet therapy is expected to counteract platelet aggregation during intravenous thrombolysis, improving the efficacy of intravenous thrombolysis as well as the functional prognosis. According to current evidence, mainstream guidelines clearly state that the administration of intravenous aspirin (or other antiplatelet agents) within 24 hours of Recombinant tissue plasminogen activator (rt-PA) thrombolytic therapy is not recommended as an adjunctive treatment of intravenous thrombolysis therapy, despite the fact that rt-PA thrombolytic therapy is still acceptable for patients who have received antiplatelet therapy before the onset of stroke. Evidence from high-quality clinical trials for the routine use of oral antiplatelet drugs before and within 24 hours of intravenous thrombolysis in acute ischemic stroke (AIS) patients is quite limited. Meanwhile, trials including INSPIRES and CHANCE 2 have demonstrated that early initiation of dual antiplatelet therapy could significantly reduce the risk of recurrence and thus improve the functional prognosis without significantly increasing the risk of bleeding, providing a promising treatment for early oral antiplatelet therapy in patients undergoing intravenous thrombolysis.

This trial is a multicenter, randomized, double-blind, placebo-parallel controlled designed clinical trial. A total of 1380 patients (aged 18-80 years) who have a new diagnosed ischemic stroke (within 6 hours of onset), a NIHSS score of 4-10 points, and have received/are planned to receive intravenous thrombolysis therapy with will be enrolled from 50 centers in China. Patients will be randomly assigned into intervention (dual antiplatelet therapy of Ticagrelor and Aspirin) and control group (placebo) by the ratio of 1:1. Face to face or distance (via video or telephone) interviews will be made at baseline, 7 ± 1 days, 30 ± 3 days, 60 ± 5 days and 90 ± 7 days after randomization.

Primary outcome is defined as good functional outcomes (mRS score of 0-1 points) at 90 days. Secondary outcomes include neurologic improvement，quality of life ( quality-of-life EuroQol-5 Dimensions scale)，activity of daily living (Barthel index)，recurrent ischemic stroke. Safety outcomes, relating to antiplatelet and intravenous thrombolysis therapy (i.e., symptomatic intracranial hemorrhage, parenchymal hematoma type 2, bleeding events) will also be investigated.

The Chi-square test was used to compare the proportion difference of good functional outcomes between two groups after 90 days of treatment, and the 95% confidence interval (CI) was calculated by using the Newcombe method. The generalized linear regression model was used to calculate the relative risk (RR) and its 95%CI. For survival outcomes, hazard ratio (HR) and 95% CI were calculated using the Cox proportional risk model.

ELIGIBILITY:
Inclusion Criteria:

* 1. 18-80 years old;

  2. Clinical diagnosis of acute ischemic stroke;

  3. Time from onset to treatment ≤6.0 hours;

  4. Having received or planning to receive intravenous thrombolytic therapy;

  5. NIHSS score of 4-10 points, and at least one of the 5th (upper limb exercise) or 6 th (lower limb exercise) scale is ≥1 point;

  6. Signed informed consent.

Exclusion Criteria:

* 1. Planning to receive endovascular therapy;

  2. mRS scores ≥2 points before the onset;

  3. Receiving any antiplatelet therapy after the onset;

  4. Bleeding or other pathological brain disorders, such as vascular malformations, tumors, abscesses, or other common non-ischemic brain diseases (such as multiple sclerosis), identified by CT/MRI;

  5. Pre-existing clotting disorders, systemic bleeding, thrombocytopenia, or neutropenia;

  6. Pre-existing atrial fibrillation or anticoagulant therapy (warfarin, heparin, thrombin inhibitors or factor Xa inhibitors);

  7. Hepatic or renal insufficiency (hepatic insufficiency refers to the alanine transaminase (ALT) value > 2 times the upper limit of normal value or aspartate aminotransferase (AST) times > 2 times the upper limit of normal value; renal insufficiency refers to creatinine values > 2 times the upper limit of normal value);

  8. Allergic to Ticagrelor or Aspirin or thier components and excipients;

  9. Women who are pregnant or breastfeeding, or those with negative pregnancy test records while refusing to use effective contraceptives;

  10. Having participated investigational drugs or device tests within 30 days;

  11. Being considered inappropriate to participate by researchers.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1382 (Actual)
Dates: Start 2024-04-03 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-01-05 (Actual)

PRIMARY OUTCOMES:
Excellent functional outcome | 90 days
  Modified Rankin Scale (mRS) score of 0-1 points; The mRS score ranges from 0 to 6, with higher scores indicating worse functional outcome.

SECONDARY OUTCOMES:
mRS score of 0-2 points | 90 days
  The mRS score ranges from 0 to 6, with higher scores indicating worse functional outcome.
Distribution of mRS score | 90 days
  The distribution of mRS score of 0 to 6 points; The mRS score ranges from 0 to 6, with higher scores indicating worse functional outcome.
Neurologic improvement | 7 days
  NIHSS score decreasing by 4 points or more than the value at baseline; The National Institutes of Health Stroke Scale (NIHSS) score ranges from 0 to 42, with higher scores indicating more severe neurological deficit.
Quality of life (EQ-5D scale) | 90 days
  The European Quality of Life 5-Dimension（EQ-5D）questionnaire for measuring generic health status. The 5-level EQ-5D version (EQ-5D-5L) comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The sum score on each of the five dimensions ranges from 5 (all domains have level 1) to 25 (all domains have level 5), with higher scores indicating worse health-related quality of life.
Activity of daily living (Barthel index ≥95 points) | 90 days
  The Barthel index score ranges from 0 to 100, with higher scores indicating greater independence.
Recurrent ischemic stroke | 90 days
Symptomatic intracranial hemorrhage (ECASS-III) | 36 hours
Symptomatic intracranial hemorrhage (ECASS-III) | 7 days
Parenchymal hematoma type 2 (SIST-MOST) | 36 hours
Parenchymal hematoma type 2 (SIST-MOST) | 7 days
Bleeding events (GUSTO) | 90 days
Adverse events | 90 days
Severe adverse events | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wang, MD, PhD, Principal Investigator — Beijing Tiantan Hospital
Locations (60):
- China (60):
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Hospital of Fangshan District, Beijing, Beijing Municipality
  - Heyuan City Hospital of Traditional Chinese Medicine, Heyuan, Guangdong
  - The Fifth Affiliated Hospital, Sun Yat-sen University, Zhuhai, Guangdong
  - Wuming Hospital of Guangxi Medical University, Nanning, Guangxi
  - Yulin First People's Hospital, Yulin, Guangxi
  - Affiliated Hospital of North China University of Science and Technology, Tangshan, Hebei
  - Linxi County People's Hospital, Xingtai, Hebei
  - Ningjin County Hospital of Hebei Province, Xingtai, Hebei
  - Qinghe People's Hospital, Xingtai, Hebei
  - Renze District People's Hospital, Xingtai, Hebei
  - Xingtai Ninth Hospital, Xingtai, Hebei
  - The First Affiliated Hospital of Hebei North University, Zhangjiakou, Hebei
  - Yangyuan County People's Hospital, Zhangjiakou, Hebei
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Puyang Anyang District Hospital, Anyang, Henan
  - Henan Wenxian People's Hospital, Jiaozuo, Henan
  - Jiaozuo People's Hospital, Jiaozuo, Henan
  - Jiyuan Hospital of Traditional Chinese Medicine, Jiyuan, Henan
  - Kaifeng Central Hospital, Kaifeng, Henan
  - Lankao County Hospital of Traditional Chinese Medicine, Kaifeng, Henan
  - Qi County Traditional Chinese Medicine Hospital, Kaifeng, Henan
  - Qixian People's Hospital, Kaifeng, Henan
  - The People's Hospital of Weishi, Kaifeng, Henan
  - Xiangfu District First People's Hospital, Kaifeng, Henan
  - Luoyang First People's Hospital, Luoyang, Henan
  - Luoyang Mengjin People's Hospital, Luoyang, Henan
  - Song County People's Hospital, Luoyang, Henan
  - Sanmenxia Hospital of the Yellow River, Affiliated to Henan University of Science and Technology, Sanmenxia, Henan
  - Henan Sui County Hospital of Traditional Chinese Medicine, Shangqiu, Henan
  - Suixian People's Hospital, Shangqiu, Henan
  - Weishi Central Hospital, Weishi Chengguanzhen, Henan
  - Weishi County Central Hospital, Weishi Chengguanzhen, Henan
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Huangpi District People's Hospital of Wuhan City, Wuhan, Hubei
  - Liuyang Jili Hospital, Changsha, Hunan
  - Chenzhou First People's Hospital, Chenzhou, Hunan
  - Chenzhou Fourth People's Hospital, Chenzhou, Hunan
  - Tuquan People's Hospital, Hinggan, Inner Mongolia
  - Zhalantun City Hospital of Chinese and Mongolian Medicine, Hulunbuir, Inner Mongolia
  - Anshan Changda Hospital, Anshan, Liaoning
  - Benxi Central Hospital, Benxi, Liaoning
  - Dalian Lvshun district people's hospital, Dalian, Liaoning
  - Dalian University Affiliated Xinhua Hospital, Dalian, Liaoning
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Dandong Central Hospital, Dandong, Liaoning
  - The First People's Hospital of Shenyang, Shenyang, Liaoning
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Neimenggu
  - Lingbao First People's Hospital, Henan, Sanmenxia
  - Yantai Penglai Traditional Chinese Medicine Hospital, Dengzhou, Shandong
  - Linyi City People Hospital, Linyi, Shandong
  - Weihai Wendeng District People's Hospital, Weihai, Shandong
  - Zibo Municipal Hospital, Zibo, Shandong
  - Yuci District People's Hospital, Jinzhong, Shanxi
  - Linfen Central Hospital, Linfen, Shanxi
  - Linfen People's Hospital, Linfen, Shanxi
  - Weinan Central Hospital, Weinan, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin Xiqing Hospital, Tianjin, Tianjin Municipality
  - The First Afflicted Hospital of Shihezi University, Shihezi, Xinjiang

REFERENCES:
- [Derived] Wang A, Xia X, Bath PM, Turc G, Li J, Zhang X, Wang Y. Rationale and design of Ticagrelor with Aspirin Dual Antiplatelet Therapy Combined with Intravenous Thrombolysis in Patients with Ischemic Stroke (TAPIS): a multicentre, randomised, double-blind, parallel group, placebo-controlled trial. Stroke Vasc Neurol. 2026 Jan 29:svn-2025-004721. doi: 10.1136/svn-2025-004721. Online ahead of print. PMID 41611343